CLINICAL TRIAL: NCT00000872
Title: Early Intensive Antiretroviral Combination Therapy in HIV-1 Infected Infants and Children
Brief Title: Treatment With Combinations of Several Antiviral Drugs in Infants and Young Children With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG 356; 10605 (Registry Identifier: DAIDS ES); PACTG 356
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; HIV-1; Drug Therapy, Combination; Zidovudine; Nevirapine; Stavudine; HIV Protease Inhibitors; CD4 Lymphocyte Count; Lamivudine; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Nelfinavir; Nevirapine; Lamivudine; Stavudine; Zidovudine

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Nelfinavir mesylate
Drug: Nevirapine
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine

SUMMARY:
This trial tests the safety and effectiveness of the early use of combinations of anti-HIV drugs in HIV-infected infants and young children in an effort to block virus growth and preserve normal immune functions.

Various anti-HIV drug combinations need to be tested in order to find the best way to treat infants and children who have been infected with HIV during birth.

DETAILED DESCRIPTION:
This study examines the antiretroviral activity of ZDV/3TC/NVP in vertically-infected infants and children aged 15 days up to 2 years, and ZDV/3TC/NVP/ABC in vertically-infected infants and children aged 30 days up to 2 years. This study will assess HIV-1 and CD4/CD8 T-cell kinetics, activation, and maturation. It will also test the concept that early (younger than 3 months of age) use of potent, combination antiretroviral therapy will allow the long-term control of viral replication with preservation of normal immune function. [AS PER AMENDMENT 3/11/98: This study will also examine the antiretroviral activity of ZDV/3TC/NVP/NFV in vertically infected infants and children.]

This is a 2-part Phase I/II, open-label trial in HIV-infected infants. Part A assesses the triple combination of ZDV, 3TC, and NVP. Four to eight patients are enrolled in each age cohort (Cohort 1: at least 15 days, no more than 3 months; Cohort 2: over 3 months, no more than 2 years). Part B assesses the quadruple combination of ZDV, 3TC, NVP, and ABC. Eight patients are enrolled in each age cohort (Cohort 3: at least 30 days, no more than 3 months; Cohort 4: over 3 months, no more than 2 years). [AS PER AMENDMENT 3/11/98: This study is now a 3-part Phase I/II trial. Parts A and B are as above. Part C will assess the quadruple regimen of d4T, 3TC, NVP and NFV. Up to 8 patients will be enrolled in each age cohort (Cohort 5: at least 15 days, no more than 3 months; Cohort 6: over 3 months, no more than 2 years). If 3 of 4 patients in either cohort of Part B do not achieve plasma RNA less than 1,000 copies/ml after 16 weeks of quadruple therapy, enrollment of patients to that cohort will stop and enrollment of 8 patients to the corresponding cohort in Part C will begin. For Part C, patients whose RNA level is no more than 1,000 copies/ml at Week 16 will remain on assigned treatment until Week 104. If at any time between Weeks 16 and 104 a patient's RNA level increases to greater than 1,000 copies/ml, plasma RNA will be repeated within 1 week. If both RNA levels are greater than 1,000 copies/ml, the patient will discontinue study treatment and be followed every 12 weeks for 1 year.] [AS PER AMENDMENT 4/14/99: The study has been extended for an additional 96 weeks for children with continued suppression of viral replication (RNA less than 400 copies/ml) at Week 104. If at any time between Week 12 or 16 and Week 200 a patient's RNA level increases to greater than 1,000 copies/ml, plasma RNA will be repeated within 1 week. If both RNA levels are above 1,000 copies/ml, the patient will discontinue treatment for best available therapy and be followed every 12 weeks for 1 year following the discontinuation of study treatment.] [AS PER AMENDMENT 9/16/99: An additional cohort (Cohort 7) of 5 to 10 patients has been added. Cohort 7 includes patients between 15 days and 3 months of age. Cohort 7 patients who experience suppression of viral replication at Week 104 are followed through Week 200.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are 15 days to 2 years old.
* Have consent of parent or legal guardian.
* Are HIV-positive.

Exclusion Criteria

Children will not be eligible for this study if they:

* Have certain infections which require treatment during the study.
* Have received certain medications.

Ages: 15 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Antiretroviral activity of ZDV/3TC/NVP | Throughout study
Durability of viral suppression | Throughout study
Immune competence and HIV-1 specific immune respones with prolonged viral suppression beyond 104 weeks | Throughout study
Antiretroviral activity of ZDV/3TC/NVP/1592U89 regimen | Throughout study
Antiretroviral activity of d4T/3TC/NVP/NFV regimen | Throughout study
Tolerance and pharmacokinetic profile of NFV | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Luzuriaga, Study Chair
Locations (12):
- United States (12):
  - Univ. of Florida College of Medicine-Dept of Peds, Div. of Immunology, Infectious Diseases & Allergy, Gainesville, Florida
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Univ. of Mississippi Med. Ctr Children's Hosp., Detroit, Michigan
  - Nyu Ny Nichd Crs, New York, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
  - Children's Hosp. of the King's Daughters, Infectious Disease, Norfolk, Virginia

REFERENCES:
- [Background] Luzuriaga K, McManus M, Britto P, Wu HL, Lindsey J, Sullivan JL. Viral kinetics and control of replication following potent early combination antiretroviral therapy of vertical HIV-1 infection. HIV Pathog Treat Conf. 1998 Mar 13-19;52 (abstract no 2024)
- [Background] Capparelli E, Sullivan J, Mofenson L, Smith B, Graham B, Britto P, Becker M, Luzuriaga K. Pharmacokinetics (PK) of nelfinavir and its metabolite (M8) in HIV-infected infants following BID or TID administration. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 729)
- [Background] Luzuriaga K, Wu H, McManus M, Britto P, Borkowsky W, Burchett S, Smith B, Mofenson L, Sullivan JL. Dynamics of human immunodeficiency virus type 1 replication in vertically infected infants. J Virol. 1999 Jan;73(1):362-7. doi: 10.1128/JVI.73.1.362-367.1999. PMID 9847340
- [Background] Luzuriaga K, Mcmanus M, Britto P, Wu H, Lindsey J, Smith B, Mofenson L, Sullivan JL. Early combination antiretroviral therapy of vertical HIV-1 infection: viral kinetics and control of viral replication. Conf Retroviruses Opportunistic Infect. 1998 Feb 1-5;5th:225 (abstract no LB12)
- [Background] Capparelli EV, Sullivan JL, Mofenson L, Smith E, Graham B, Britto P, Becker MI, Holland D, Connor JD, Luzuriaga K; Pediatric ACTG 356 Investigators. Pharmacokinetics of nelfinavir in human immunodeficiency virus-infected infants. Pediatr Infect Dis J. 2001 Aug;20(8):746-51. doi: 10.1097/00006454-200108000-00006. PMID 11734735
- [Background] Luzuriaga K, McManus M, Mofenson L, Britto P, Graham B, Sullivan JL; PACTG 356 Investigators. A trial of three antiretroviral regimens in HIV-1-infected children. N Engl J Med. 2004 Jun 10;350(24):2471-80. doi: 10.1056/NEJMoa032706. PMID 15190139
- [Derived] McManus M, Henderson J, Gautam A, Brody R, Weiss ER, Persaud D, Mick E, Luzuriaga K; PACTG 356 Investigators. Quantitative Human Immunodeficiency Virus (HIV)-1 Antibodies Correlate With Plasma HIV-1 RNA and Cell-associated DNA Levels in Children on Antiretroviral Therapy. Clin Infect Dis. 2019 May 2;68(10):1725-1732. doi: 10.1093/cid/ciy753. PMID 30668843